CLINICAL TRIAL: NCT04476953
Title: COVID-FISETIN: A Phase 2 Placebo-Controlled Pilot Study in SARS-CoV-2 of Fisetin to Alleviate Dysfunction and Excessive Inflammatory Response in Hospitalized Adults
Brief Title: COVID-FISETIN: Pilot in SARS-CoV-2 of Fisetin to Alleviate Dysfunction and Inflammation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Paschalis Vergidis, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-003936
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Covid19
Keywords: SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — fisetin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): Subjects will receive treatment drug Fisetin
  Interventions: Drug: Fisetin
- Placebo Group (Placebo Comparator): Subjects will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo looks exactly like the study drug, but it contains no active ingredient.
  Arms: Placebo Group
Drug: Fisetin — ~20 mg/kg/day oral, NG or D tube course for 2 consecutive days
  Other Names: 3,3',4',7-tetrahydroxyflavone
  Arms: Treatment Group

SUMMARY:
The purpose of this study is to test whether Fisetin, a senolytic drug, can assist in preventing an increase in the disease's progression and alleviate complications of coronavirus due to an excessive inflammatory reaction.

DETAILED DESCRIPTION:
To determine if Fisetin treatment can prevent deterioration of oxygenation status as measured by S/F ratio: SpO2/ FiO2, as well as prevent deterioration in physical function (frailty) and hyper-inflammation, other measures of oxygenation status (progression to supplemental oxygen requirement, assisted breathing/ ventilation), and progression from mild/ moderate to severe/ critical proven SARS-CoV-2 infection in hospitalized patients and to evaluate the safety and tolerability of Fisetin in this patient population.

ELIGIBILITY:
Inclusion Criteria - Patients must meet all of the following inclusion criteria to be enrolled in this study.

1. Men or women 60 years of age or older

   OR

   Age 18 - 59 years WITH at least one of the following comorbidities:
   * BMI greater than or equal to 35
   * Diabetes
   * Asthma/ Chronic Obstructive Pulmonary Disease (COPD)
   * Previous Myocardial Infarction
   * Previous Stroke/ Cerebrovascular Accident (CVA)
   * Hypertension/ Atherosclerosis/ Peripheral Vascular Disease
   * Smoking and/or vaping
   * Other conditions associated with senescent cell accumulation (i.e. previous chemotherapy or radiation)
2. SpO2 greater than or equal to 85% (on room air or less than or equal to 2 L of supplemental oxygen)
3. Willing and able to provide written informed consent or have a legally authorized representative (LAR) who will provide informed consent
4. SARS-CoV-2 infection confirmed by PCR test at Mayo Clinic (or other CLIA certified) laboratory within 10 days prior to randomization.

Exclusion Criteria - Patients who meet any of the following exclusion criteria are not to be enrolled in this study.

General Exclusion Criteria

1. Presence of any condition that the Investigator or the subject's attending physician believes would put the subject at risk or would preclude the patient from successfully completing the trial
2. Pregnant and/or lactating. Women of childbearing potential (WCBP) must have a negative pregnancy test within 72 hours prior to randomization
3. WCBP who are unwilling to abstain from sex or use an adequate method of contraception from the time of the first IP administration through 48 hours after the last IP administration
4. Men who are unwilling to abstain from sex with WCBP or use an adequate method of contraception from the time of the first IP administration through 48 hours after the last IP administration

   Laboratory Exclusion Criteria
5. Total bilirubin >3X upper limit of normal or as per clinical judgment.
6. Serum aspartate transaminase (AST) or alanine aminotransferase (ALT) >4x the upper limits of normal or as per clinical judgment.
7. Hemoglobin <7 g/dL; white blood cell count ≤ 2,000/mm3 (< or = 2.0 x 109/L) or > or = 20,000/mm3 (> or = 20 x 109/L); platelet count < or = 40,000/µL (< or = 40 x 109/L); absolute neutrophil count < or = 1 x 109/L; lymphocyte count <0.3 x 109/L at screening or as per clinical judgment.
8. Unstable (as per clinical judgment) major cardiovascular, renal, endocrine, immunological, or hepatic disorder.
9. eGFR <25 ml/ min/ 1.73 m2 or as per clinical judgment.
10. Plasma and/or serum glucose >300 or as per clinical judgment.

    Clinical History Exclusion Criteria
11. Human immunodeficiency virus infection.
12. Known active hepatitis B or C infection.
13. Invasive fungal infection.
14. Uncontrolled (as per clinical judgement) pleural/pericardial effusions or ascites.
15. New/active invasive cancer except non-melanoma skin cancers.

    Medication Exclusion Criteria (See Appendices 1-3 for additional information)
16. Known hypersensitivity or allergy to Fisetin.
17. Patients currently using medications which utilize CYP450 2C9 for metabolism. These medications include: Fosphenytoin, Phenytoin, Warfarin, Glimepiride, Diclofenac, Bosentan, and Glyburide. Patients taking any of these medications may participate if the medications can be held immediately before the 1st IP administration until at least 10 hours after the last (2nd) IP administration and the patient is otherwise eligible.
18. Patients currently using medications which utilize CYP2C9, CYP2C19, CYP1A2, OATP1B1. These medications include: Olanzapine, Clozapine, Theophylline, Tizanidine, Warfarin, Rameltoen, Tacrine, Duloxetine, Mexiletine, Riluzole, and Atomoxetine. Patients taking any of these medications may participate if the medications can be held immediately before the 1st IP administration until at least 10 hours after the last (2nd) IP administration and the patient is otherwise eligible.
19. Patients currently using medications which are strong inhibitors of CYP3A4. These medications include: Atazanavir, Ceritinib, Clarithromycin, Darunavir, Idelalisib, Indinavir, Itraconazole, Ketoconazole, Lopinavir, Mefipristone, Nefazodone, Nelfinavir, Ombitasivir-paritaprevir-ritonivir, Ombitasivir-paritaprevir-ritonivir-plus dasabuvir, Posaconazole, Saquinavir, Telithromycin, Tucatinib, and Voriconazole. Patients taking any of these medications may participate if the medications can be held immediately before the 1st IP administration until at least 10 hours after the last (2nd) IP administration and the patient is otherwise eligible.
20. Patients currently using antifungals. If antifungals are absolutely necessary from an infectious disease perspective, then they will be allowed only if the levels are subtherapeutic or therapeutic.
21. Patients taking any of these medications may participate if the medications can be held immediately before the 1st IP administration until at least 10 hours after the last (2nd) IP administration and the patient is otherwise eligible:

    * Cardiac: digoxin, flecainide, amiodarone
    * Psychiatric: lithium, thioridazine
    * Neurologic: carbamazepine, phenobarbital
    * Antimicrobial/fungal: aminoglycosides (e.g. amikacin, gentamicin, kanamycin, neomycin, netilmicin, paromomysin, streptomycin, tobramycin), rifampin
    * Anticoagulants/ Antiplatelets: warfarin
    * Others: methotrexate, nitroglycerin, St. John's wort, tyrosine kinase inhibitors, tacrine, diclofenac
22. Participation in other clinical trials involving treatment for SARS-CoV-2. (unless reviewed and approved by the Principal Investigator). Note that institutional standard of care treatment of SARS-CoV-2 including glucocorticoids, hydroxychloroquine, azithromycin, remdesivir, anti-spike antibodies, and/or convalescent plasma are not excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events | 6 months
  Number of participants to experience serious adverse events and hypersensitivity reactions.
Change in oxygenation status | baseline, Day 3, 7, 10, 14, 17 and 30; Months 3 and 6
  change in oxygenation levels as measured by S/F ratio (SPO2/FiO2)

SECONDARY OUTCOMES:
CoV Severity Category | 6 months
  Number of participants to progress to severe or critical classification CoV

CONTACTS AND LOCATIONS:
Overall Officials: Paschalis Vergidis, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No